CLINICAL TRIAL: NCT04537481
Title: Lipidic Profiles Differences of Sperm Between Normal and Low Fertilization Male Patients in Vitro Fertilization
Brief Title: Lipidic Differences of Sperm Between Normal and Low Fertilization Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: L0805
Record Dates: First submitted 2020-08-19; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Fertilization
Keywords: In vitro fertilization (IVF); Sperm; Fertilization; Lipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal fertilization group (Experimental): Sperm samples from the successful fertilization IVF cycles were collected.
  Interventions: Other: Lipid extraction
- Low fertilization group (Experimental): Sperm samples from the low fertilization IVF cycles were collected.
  Interventions: Other: Lipid extraction

INTERVENTIONS:
Other: Lipid extraction — The sperm samples were used for lipid extraction. Lipids were analyzed using the UPLC-MS system.

SUMMARY:
Although in vitro fertilization (IVF) involve the use of semen samples, there is little scientific methodology applied when selecting sperm. To select the most appropriate spermatozoa, first the operator need to define the optimal molecular markers. Sperm lipids may contribute to sperm function, thus the investigator's aim was to compare the lipidic profiles differences of sperm samples used in IVF cycles that ultimately led to normal fertilization or low fertilization.

DETAILED DESCRIPTION:
There is increasing evidence that male fertility/infertility and sperm physiology are determined by multiple factors, necessitating the use of numerous molecular biomarkers to precisely assess male reproductive potential. The study has reported that the lipids are special interest as fertility markers and therapeutic targets not only due to their functions in sperm, but also because they are sensitive to external and environmental signals.

Sperm samples from infertile patients after IVF ( normal fertilization group, n=25; low fertilization group, n=25) were collected. Following standard density gradient separation operating procedure, the sample were incubated in 37°C, 5%CO2, for 3 hours. The sample included 10x10^6 spermatozoa after sample preparation and aliquots in 100 μL PBS were analyzed for lipid composition using ultra-high performance liquid chromatography coupled to mass spectrometry. Lipid compositions and levels were compared between the two groups. The results will describe the composition and contents of lipids linked to capacitation of sperm, opening a new possibilities for the development of male fertility diagnostic tools and culture media formulations to improve sperm quality and enhance fertilization result.

ELIGIBILITY:
Inclusion Criteria:

* Tubal factor infertility,
* The women's BMI (Body mass index) ranged from 18.5 to 24,
* The women's AMH (Anti-Müllerian hormone) ranged from 2 to 6.8 ng/ml,
* The oocyte mature rate was greater than 75%,
* 8 ≤ Number of retrieved oocytes ≤ 16.
* Analysis of the spouse's semen conventional parameters showed normal.

Exclusion Criteria:

* The age is over 35 years old.
* The women with polycystic ovary syndrome (PCOS).
* The endocrine function of the women was disordered.
* The women has metabolic disease.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Normal fertilization rate | 6 months
  2PN (two pronuclei and two polar bodies) rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Bo, Doctor, Study Chair — Reproductive Medicine Center, Tangdu Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No